CLINICAL TRIAL: NCT02933229
Title: The Influence of Helicobacter Pylori Eradication on Gastric Pathology: a Long-term, Prospective Cohort Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016SDU-QILU-19
Record Dates: First submitted 2016-10-11; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Helicobacter Pylori; the Operative Link on Gastric Intestinal Metaplasia; Operative Link on Gastric Intestinal Assessment
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- H. pylori eradication cohort (Experimental): H. pylori eradication therapy comprising esomeprazole, amoxicillin,clarithromycin and colloidal bismuth pectin.
  If failed in eradicating H. pylori, a culture based antimicrobial susceptibility test will be used to guide H. pylori eradication.
  Interventions: Device: biopsy; Drug: H. pylori eradication

INTERVENTIONS:
Device: biopsy — patients enrolled in the study will receive gastroscopy and biopsies in order to evaluate status of pathology.
Drug: H. pylori eradication — H. pylori eradication therapy comprising esomeprazole, amoxicillin,clarithromycin and colloidal bismuth pectin.
  If failed in eradicating H. pylori, a culture based antimicrobial susceptibility test will be used to guide H. pylori eradication.

SUMMARY:
Helicobacter pylori (H. pylori) infection, affecting an estimated 50% of the global population, is a main cause of chronic gastritis, peptic ulcers and gastric cancer. By causing progressive damage to the stomach and may eventually result in gastric atrophy, H. pylori infection has been demonstrated to be responsible for more than 95% of gastric malignancies

ELIGIBILITY:
Inclusion Criteria:

* Patients with H. pylori infection;
* Aged 18-65 years.

Exclusion Criteria:

* Patients with gastrectomy, acute GI bleeding and advanced gastric cancer;
* Conditions unsuitable for performance of gastroscopy, such as coagulopathy, impaired renal function;
* Pregnancy or breastfeeding;
* Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-10; Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of more severe inflammation in the gastric mucosa for 15 years after H. pylori eradication at five points of the stomach compared with original status | 15 years
The proportion of more severe atrophy in the gastric mucosa for 15 years after H. pylori eradication at five points of the stomach compared with original status | 15 years
The proportion of more severe IM in the gastric mucosa for 15 years after H. pylori eradication at five points of the stomach compared with original status | 15 years

SECONDARY OUTCOMES:
The proportion of more advanced stages for 15 years after H. pylori eradication by using operative link on gastritis assessment (OLGA) system compared with original status. | 15 years
The proportion of more advanced stages for 15 years after H. pylori eradication by using operative link for gastritis intestinal metaplasia (OLGIM) system compared with original status. | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Li Yanqing, MD, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No